CLINICAL TRIAL: NCT02060565
Title: Prognosis Value of Non-invasive Methods for the Diagnosis of Chronic Liver Disease. a Retrospective and Prospective 20-year Follow-up.
Brief Title: Prognosis Value of Non-invasive Methods for the Diagnosis of Chronic Liver Disease
Acronym: PVNIM
Status: Recruiting | Type: Observational
Sponsor: Association HGE CHU Bordeaux Sud (Other)
Responsible Party: Sponsor
Other Study IDs: HL V-0214
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Chronic Liver Disease
Keywords: diagnosis; survival; non-invasive method; cirrhosis; FibroScan
MeSH Terms: conditions — Disease; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic liver disease: all patients with chronic liver disease followed using non-invasive methods

SUMMARY:
The aim of this retrospective and prospective study is to evaluate the 20-year prognosis value of non-invasive methods for the diagnosis of chronic liver disease for predicting survival and complications of cirrhosis.

DETAILED DESCRIPTION:
All consecutive patients with chronic liver disease will be followed during 20 years.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C
* chronic hepatitis B
* alcohol liver disease
* non alcoholic liver disease

Exclusion Criteria:

* ascitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients with an age over eighteen and chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 20 years

SECONDARY OUTCOMES:
Survival without liver complications | 20 years

OTHER OUTCOMES:
Survival without liver transplantation | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Foucher, MD, Study Chair — Association HGE CHU Bordeaux Sud; Faiza Chermak, MD, Study Chair — Association HGE CHU Bordeaux Sud; Victor de Lédinghen, MD, PhD, Study Director — Association HGE CHU Bordeaux Sud; Jean-Baptiste Hiriart, MD, Study Chair — Association HGE CHU Bordeaux Sud
Locations (1):
- Centre d'Investigation de la Fibrose hépatique Service Hépato-Gastroentérologie Hopital Haut-Lévèque, Pessac, France